CLINICAL TRIAL: NCT06205823
Title: A Retrospective Study to Compare Clinical Outcomes Between Advanced Immunotherapy and Classical Immunochemotherapy in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Compare Clinical Outcomes Between Advanced Immunotherapy and Classical Immunochemotherapy in RRMM
Acronym: CAREMM-2305
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Sung-Soo Park, Principal Investigator, Seoul St. Mary's Hospital
Other Study IDs: XC23RIDI0066
Record Dates: First submitted 2023-12-17; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Myeloma Multiple
MeSH Terms: conditions — Multiple Myeloma | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T cell engager
  Interventions: Drug: Immunotherapy
- Standard-of-care
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — Immunotherapy

SUMMARY:
[Purpose]

This study aims to assess the efficacy of immunotherapeutic agents in real clinical settings by comparing the treatment outcomes of relapsed/refractory multiple myeloma patients treated with immunotherapeutic agents and classical immunotherapeutic agents.

[Primary Study Objective] Compare the overall survival duration among patients based on the administered treatments.

[Secondary Study Objectives] Compare the progression-free survival duration among patients based on the administered treatments.

Compare the response rates among patients based on the administered treatments. Compare the healthcare costs associated with the administered treatments among patients.

[Study Participants]

Patients diagnosed with plasma cell disorders (PCD) at Seoul St. Mary's Hospital, Yeouido St. Mary's Hospital, Incheon St. Mary's Hospital, and Eunpyeong St. Mary's Hospital from May 2009 to June 2023.

- Selection Criteria

1. Patients diagnosed with multiple myeloma at Seoul St. Mary's Hospital, Yeouido St. Mary's Hospital, Incheon St. Mary's Hospital, and Eunpyeong St. Mary's Hospital from May 2009 to June 2023.
2. Age 19 and above.
3. Patients who have undergone immunotherapy* for the purpose of treating relapsed/refractory multiple myeloma.

   *Immunotherapy is defined as one of the following drugs depending on the treatment timeline:Proteasome inhibitor, immune modulatory drug, monoclonal antibody, Chimeric Antigen Receptor T-cell therapy (CAR-T), bispecific antibody, antibody-drug conjugate.
4. Exclusion Criteria:

   Patients diagnosed with conditions other than monoclonal gammopathy of undetermined significance (MGUS) or multiple myeloma.
5. Data Collection Period for Study Participants : April 1, 2009, to June 30, 2023.

[ Study plan] This study is a cross-sectional study that includes all patients who meet the selection criteria for a specific period.

All participants meeting the selection criteria are included in the study and investigated for the items.

Among the study participants, patients who received immunotherapy agents defined as immune checkpoint inhibitors are identified as the experimental group.

The entire cohort is initially defined as the control group for the experimental group.

From the initial control group, a final control group is determined by matching with the experimental group based on specific variables, including treatment cycles, in a 1:4 ratio. However, the cohort size for matching can be adjusted during the study. Comparative analyses are conducted between the experimental and control groups, examining baseline variables and outcome variables.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with multiple myeloma at Seoul St. Mary's Hospital, Yeouido St. Mary's Hospital, Incheon St. Mary's Hospital, and Eunpyeong St. Mary's Hospital from May 2009 to June 2023.
2. Age 19 and above.
3. Patients who have undergone immunotherapy* for the purpose of treating relapsed/refractory multiple myeloma.

   * Immunotherapy is defined as one of the following drugs depending on the treatment timeline:

Proteasome inhibitor, immune modulatory drug, monoclonal antibody, Chimeric Antigen Receptor T-cell therapy (CAR-T), bispecific antibody, antibody-drug conjugate.

Exclusion Criteria:

* Patients diagnosed with conditions other than monoclonal gammopathy of undetermined significance (MGUS) or multiple myeloma.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with plasma cell disorders (PCD) at Seoul St. Mary's Hospital, Yeouido St. Mary's Hospital, Incheon St. Mary's Hospital, and Eunpyeong St. Mary's Hospital from May 2009 to June 2023.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of Survival Periods Among Groups Comparison of Survival Periods Among Groups | Up to 2 years
  overall survival

SECONDARY OUTCOMES:
Comparison of Progression-Free Survival Periods | Up to 2 years
  progression-free survival
Comparison of Response Rates | Up to 2 years
  response rate
Cost-effectiveness measured by incremental Cost-effectiveness ratio (ICER) | Up to 2 years
  cost-effectiveness ratio

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Soo Park, Dr., Study Director — Seoul
Locations (1):
- Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi S, Byun JM, Park SS, Han J, Oh S, Jung S, Park H, Han S, Lee JY, Koh Y, Jeon YW, Yahng SA, Shin SH, Yoon SS, Min CK. Efficacy and Safety of Bispecific T-Cell Engagers in Relapsed/Refractory Multiple Myeloma: A Real-World Data-Based Case-Controlled Study. Transplant Cell Ther. 2025 Feb;31(2):74.e1-74.e11. doi: 10.1016/j.jtct.2024.11.010. Epub 2024 Nov 26. PMID 39608453